CLINICAL TRIAL: NCT03226132
Title: Biobehavioral Mechanisms Underlying Improving Sleep to Reduce Risk for Substance Use Disorder
Brief Title: Improving Sleep to Reduce Risk for Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Short01
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Substance Use Disorders; Insomnia; Posttraumatic Stress Disorder
MeSH Terms: conditions — Substance-Related Disorders; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Treatment for Insomnia (Experimental): Brief Behavioral Treatment for Insomnia
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia
- Repeated Contact (Active Comparator): Repeated Contact
  Interventions: Behavioral: Repeated Contact

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia — Brief Behavioral Therapy for Insomnia
  Arms: Brief Behavioral Treatment for Insomnia
Behavioral: Repeated Contact — Repeated Contact
  Arms: Repeated Contact

SUMMARY:
Substance use disorders (SUDs) are a prevalent and impairing condition, particularly among trauma exposed individuals. The current proposal aims to address the critical need for targeted direct SUD prevention in this population by intervening on a novel, malleable risk factor for SUD common among trauma-exposed individuals: sleep disturbance. Sleep disturbance prospectively predicts the development of SUD and may confer risk for SUD by increasing stress reactivity, decreasing decision-making abilities, and ultimately promoting substance use to relieve negative affect, a core etiological factor in SUD. However, to our knowledge, no experimental studies have determined whether improving sleep leads to reductions in SUD risk. As such, the current study will use a randomized controlled trial design to test the effects of brief behavioral treatment for insomnia (BBTI) against a waitlist control among a sample of trauma-exposed young adults with poor sleep and risk for SUD (N = 60). We aim to determine the direct and indirect effects of condition (BBTI vs. waitlist control) on SUD symptoms, substance use-related problems, coping motives, and posttraumatic stress symptoms through improvements in sleep. Furthermore, we will test direct and indirect effects of condition on theoretically proposed mechanisms underlying the association between sleep disturbance and SUD risk (i.e., stress reactivity, cravings in response to stress).

ELIGIBILITY:
Inclusion Criteria:

* Trauma exposure
* Current cannabis use
* Insomnia symptoms
* Age 18-30

Exclusion Criteria:

* Severe substance use disorder
* Receiving treatment related to sleep or substance use

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from Baseline to Three Months Follow-Up
PTSD Symptoms (PTSD Checklist-5) | Change from Baseline to Three Months Follow-Up
Substance Use Disorder Symptoms (Cannabis Use Disorder Identification Test; Structured Clinical Interview for Diagnostic and Statistical Manual [DSM]-5) | Change from Baseline to Three Months Follow-Up
Substance Use Motives (Marijuana Motives Measure) | Change from Baseline to Three Months Follow-Up
Substance Use Frequency (Timeline Followback) | Change from Baseline to Three Months Follow-Up

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No